CLINICAL TRIAL: NCT02226952
Title: A Randomised, Double-blind, Placebo Controlled Trial With 25 mg, 200 mg and 500 mg BILN 2061 ZW Given p.o. at Two Consecutive Days Bid to Investigate the Antiviral Efficacy, Pharmacokinetics, Safety in Patients With Chronic Hepatitis C Virus Infection
Brief Title: Antiviral Efficacy, Pharmacokinetics and Safety of BILN 2061 ZW in Patients With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 605.5
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (6):
- Group 1 (Experimental): BILN 2061 W, medium dose, in patients with genotype 1, minimal fibrosis
  Interventions: Drug: BILN 2061 W, medium dose
- Group 2 (Experimental): BILN 2061 W, high dose, in patients with genotype 1, minimal fibrosis
  Interventions: Drug: BILN 2061 W, high dose
- Group 3 (Experimental): BILN 2061 W, high dose, in non-genotype 1 patients, minimal fibrosis
  Interventions: Drug: BILN 2061 W, high dose
- Group 4 (Experimental): BILN 2061 W, low dose, in patients with genotype 1, minimal fibrosis
  Interventions: Drug: BILN 2061 W, low dose
- Group 5 (Experimental): BILN 2061 W, medium dose, in patients with genotype 1, advanced fibrosis
  Interventions: Drug: BILN 2061 W, medium dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BILN 2061 W, low dose
  Arms: Group 4
Drug: BILN 2061 W, medium dose
  Arms: Group 1; Group 5
Drug: BILN 2061 W, high dose
  Arms: Group 2; Group 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the antiviral efficacy, pharmacokinetics and tolerability of BILN 2061 ZW in a polyethyleneglycol 400 (PEG 400: ethanol) drinking solution given for two days bid in patients with chronic Hepatitis C Virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Female or male sex, age of 18 years or older
* Active, chronic Hepatitis C virus (HCV) infection
* Liver biopsy consistent with active HCV infection obtained within the last 12 months
* Written informed consent consistent with International Committee on Harmonization (ICH) / Good Clinical Practice (GCP) and local legislation given prior to any study procedures
* HCV of genotype I (Group 1, 2, 4 and 5) and non-genotype 1 (Group 3)
* HCV load greater than 50,000 copies messenger ribonucleic acid (mRNA) per ml serum at screening
* For Group 5 only: Histology showing moderate or severe fibrosis (portal fibrosis, septae, periportal and porto-central septae), no regenerative nodes and no incomplete or complete cirrhosis, corresponding to Ishak score 3 or 4, or Metavir F2 or F3 (if Ishak is not 5)

Exclusion Criteria:

* Women of childbearing potential or breastfeeding women. Postmenopausal women less than 6 months after last menses, surgically sterilized or hysterectomised patients less than 3 months after operation or without a negative serum pregnancy test
* Males not using an adequate form of contraception (condom, sterilisation at least 6 months post operation) if their partner is of childbearing potential (criteria see above) and is not using an adequate form of contraception (hormonal contraceptives, oral or injectable/ implantable, intra-uterine device (IUD))
* Any other or additional plausible cause for chronic liver disease, including the presence of other viruses known or suspected to cause hepatitis
* Ascites or other current evidence of portal hypertension
* Histology showing signs of bridging or higher grade fibrosis (e.g. Fibrosis >= Grade 3 (Ishak score) or >= 2 (Metavir score) for treatment groups 1, 2, 3, 4 or for Treatment group 5: Histology showing less than moderate or severe fibrosis (portal fibrosis, septae, periportal and porto-central septae), or showing regenerative nodes or incomplete or complete cirrhosis, corresponding to other Ishak scores than 3 or 4 and to other Metavir scores than F2 or F3 (or F3 and Ishak 5)
* History of abuse of alcohol within the past twelve months
* Planned or concurrent usage of any other pharmacological therapy at screening, including any antiviral therapy
* Any concurrent infectious disease requiring antimicrobial treatment
* History of malignancy (except for previously cured squamous cell or basal cell carcinoma)
* Usage of any investigational drug within thirty (30) days prior to enrolment; or the planned usage of an investigational drug during the course of the current study
* Known hypersensitivity to drugs
* Inability to comply with the protocol
* Prior randomization into this trial
* Child´s B or C liver diseases at screening (treatment groups 1, 2, 3, 4). Applicable for treatment group 5 only:

  * For Bilirubin - refer to following exclusion criterion
  * Quick (Prothrombin time) < 70%
  * Albumin < 3.5 g/dl
  * Clinical evidence of ascites
  * Clinical evidence of encephalopathy
* Clinically apparent jaundice or a total bilirubin or alkaline phosphatase (AP) exceeding 1.5 x upper limit of normal (ULN) at screening (treatment groups 1, 2, 3, 4). Treatment group 5 (BILN 2061 ZW, 200 mg bid/2 days in patients with advanced liver fibrosis): Clinically apparent jaundice or a bilirubin >= 2.0 mg/dl at screening. Increased alkaline phosphatase (AP) is allowed.
* ALT or AST > 5 x ULN at screening (treatment groups 1, 2, 3, 4). Treatment group 5: ALT or AST >= 10 x ULN at screening
* A platelet count of less than 100.000 platelets per mm3 at screening
* White blood cell count of less than 2,000 cells per mm3 at screening
* Positive test for human immunodeficiency Virus (HIV) at screening
* Positive test for illicit or unprescribed drugs or medications at screening. Positive test for cannabis may be allowed if the investigator assesses this result not as clinically significant
* Patients with any clinically significant laboratory abnormalities based on the investigator's medical assessment at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-11; Primary Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Virus load (VL) determined by number of copies of HCV mRNA per ml serum | up to day 14
  Cobas Amplicor HCV Monitor v 2.0 (HCM-2.0, Roche Diagnostics)

SECONDARY OUTCOMES:
Number of patients with clinically relevant changes in alanine aminotransferase (ALT) | up to day 14
Number of patients with clinically relevant changes in aspartate aminotransferase (AST) | up to day 14
Number of patients with clinically relevant changes in vital signs | up to day 14
  pulse rate, systolic and diastolic blood pressure
Number of patients with clinically relevant changes in electrocardiography (ECG) | up to day 14
Number of patients with clinically relevant changes in routine laboratory tests | up to day 14
Number of patients with adverse events | up to 35 days
Maximum concentration in plasma after a single dose administration (Cmax) | up to day 4
Area under the plasma concentration-time curve from t = 0 to t = .τ rate (AUC0-τ) | up to day 4
Time to reach Cmax following a single dose administration (tmax) | up to day 4
Total oral clearance of drug from plasma after oral administration, divided by F (CL/F) | up to day 4
Apparent volume of distribution during the terminal elimination phase (Vz/F) | up to day 4
Assessment of tolerability by investigator on a 4-point scale | day 3